CLINICAL TRIAL: NCT06403644
Title: Evaluating the Technology and Assessing the Biological Effects of Commercially Available PhotoBioModulation Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Air Force Research Laboratory (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); The Geneva Foundation (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Jason Eckerle, Principal Investigator, United States Air Force Research Laboratory
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FWR20230189H
Record Dates: First submitted 2024-03-22; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Physiological Wellness
Keywords: Photobiomodulation; Recovery; Wellness

STUDY DESIGN:
Intervention Model Description: Participants will have two 3-week periods of treatment with a washout week in-between treatment. Participants will be randomized to either sham PBM treatment or active PBM treatment first.
Who Masked: Participant
Masking Description: To prevent possible bias between the sham and active conditions, both groups will receive light filtering glasses (to control for light perception), noise-cancelling headphones, and be in a controlled temperature room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Photobiomodulation Full Body Light Bed Therapy (Active Comparator): Active treatment will be provided via a specialized full body light bed equipped with light-emitting diodes (LEDs) emitting specific wavelengths of light. The participant will be asked to lay in the bed for a 20-minute session. Treatment will be provided 3 times a week for 3 weeks.
  Interventions: Device: NovoTHOR XL Photobiomodulation Full Body Light Bed; Device: ARRC LED Photobiomodulation Full Body Light Bed
- Sham Photobiomodulation Full Body Light Bed Therapy (Sham Comparator): Sham-PBMT will be delivered in the same manner as indicated for the Active treatment process, but the devices will not be turned on. The participant will be asked to lay in a specialized full body light bed equipped with light-emitting diodes (LEDs) for a 20-minute session. Sham-PBMT Treatment will be provided 3 times a week for 3 weeks.
  Interventions: Device: NovoTHOR XL Photobiomodulation Full Body Light Bed; Device: ARRC LED Photobiomodulation Full Body Light Bed

INTERVENTIONS:
Device: NovoTHOR XL Photobiomodulation Full Body Light Bed — Low powered full-body photobiomodulation light bed therapy will be administered via the NovoTHOR XL light therapy bed which emits an average irradiance of ~30 mW/cm^2.
Device: ARRC LED Photobiomodulation Full Body Light Bed — High powered full-body photobiomodulation light bed therapy will be administered via the ARRC LED light therapy bed which emits an average irradiance of ~75 mW/cm^2.

SUMMARY:
Photobiomodulation therapy (PBMT) involves applying non-ionizing forms of light from sources including lasers, LEDs, and broadband light, in the visible and near infrared spectrum, to the body to enhance performance, stimulate healing, modulate recovery, and improve health. The investigators will conduct a single-blinded randomized-control trial with sham control to investigate the effectiveness of providing PBMT in a military population, translating this cutting-edge research to application in the operational setting.

DETAILED DESCRIPTION:
In addition to assessing the efficacy of whole-body PBMT in comparison to sham therapy, the human subjects PBM study conducted encompasses a comprehensive data collection endeavor aimed at evaluating PBMT's impact on general wellness. Using a single-blinded randomized control trial design, participants are assigned to different treatment groups and subjected to PBMT or sham treatments over specified periods. Randomization ensures unbiased assignment to treatment groups, and participants are blinded to their assigned study arm until the conclusion of the final study visit. Detailed treatment protocols are followed, including precautions to minimize bias between active and sham treatments. Data collection includes an extensive array of both subjective and physiological measures, encompassing tools such as the Defense and Veteran's Pain Rating Scale (DVPRS), Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), heart rate monitors, blood samples, and saliva samples. Additionally, this study investigates the differences between high-power PBMT (~70mW/cm2) and low-power PBMT (~30mW/cm2) by a secondary randomization of participants into one of two commercial PBMT light beds (either the NovoTHOR or ARRC LED).

The study is conducted over an 8-week period and separated into two arms. Participants that meet final eligibility criteria will be randomized to a study arm following informed consent using a computer-generated randomization model. Participants will first be randomized (1:1) to a high-power PBM (ARRC-LED) or low-power PBM (NovoTHOR) treatment group. Then participants will subsequently be randomized (1:1) to a treatment schedule (either sham or active treatment first). The initial week of the study consists of a washout week in which baseline data is collected. In Part 1 (Weeks 2-4), participants undergo photobiomodulation treatment sessions or sham photobiomodulation treatment sessions lasting 20 minutes, occurring 3 times a week for 3 weeks. Following Part 1, Week 5 consists of an additional washout period. During this 1-week period, participants will continue daily study procedures, including questionnaires, saliva collection, and wearing the Oura Ring, but will not receive sham or active PBMT. In Part 2 (Weeks 6-8), participants will resume treatment sessions crossing over into the other condition (either sham or active PBMT), also lasting 20 minutes and occurring 3 times a week for 3 weeks. Overall, the human subjects experiment works to provide valuable insights into the practical applications and potential benefits of PBMT.

ELIGIBILITY:
Inclusion Criteria:

1. Active-duty military personnel, government civilians, and government contractors
2. Between the ages of 18-45 years old (inclusive)
3. Ability to read and understand English language
4. Willingness and ability to commit to study procedures, including study intervention and follow-up

Exclusion Criteria:

1. Body fat > 40%
2. Weight exceeds 300lbs
3. Height exceeds 7ft 3in
4. > 10% of full body coverage of tattoos
5. Cardiovascular disease requiring medical management
6. Currently utilizing a pacemaker
7. Currently utilizing select medications (e.g., statins, diuretics, antihypertensive agents)
8. Currently utilizing medications associated with sensitivity to heat or light (e.g., amiodarone, chlorpromazine, doxycycline, hydrochlorothiazide, nalidixic acid, naproxen, piroxicam, tetracycline, thioridazine, voriconazole)
9. Currently undergoing treatment for a brain-related injury
10. Diagnosis of autoimmune diseases
11. Diagnosis of porphyria (light induced allergy) or photosensitive eczema
12. Diagnosis of Cancer
13. Diagnosis of epilepsy and/or being seizure prone
14. Diagnosis of diabetes
15. Diagnosis of Lupus Erythematosus
16. Diagnosis of retinal disease
17. Uncontrolled thyroid disease (known problem with no medical management)
18. Cirrhosis of the liver
19. Impaired blood clotting (from medication or underlying condition)
20. Photophobia
21. Albinism/achromasia
22. Currently pregnant or plan to become pregnant during the study (6 weeks)
23. Currently participating in any other intervention-based research studies other than protocol FWR20220097H that may confound results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2028-03-11 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Effects of PBMT versus Sham PBMT on Proinflammatory Blood Biomarkers | Through study completion, an average of 8 weeks.
  Changes in blood biomarkers (MSD proinflammatory panel: IL-1beta, IL-2, IL-6, IL-12p70, IL-17A, IFN-gamma, and TNF-alpha) compared across the sham and active PBMT conditions. As elevated proinflammatory cytokine levels may be a sign of heightened inflammation, lower proinflammatory cytokine levels at the end of the active condition compared to the beginning of the block, along with no statistical change at the end of the sham block condition compared to the beginning of the sham block, may indicate a more ideal treatment outcome.
Effects of PBMT versus Sham PBMT on Anti-Inflammatory Blood Biomarkers | Through study completion, an average of 8 weeks.
  Changes in blood biomarkers (MSD anti-inflammatory panel: IL-4, IL-10) compared across the sham and active PBMT conditions. As elevated anti-inflammatory cytokine levels may be a sign of lowered inflammation, higher anti-inflammatory cytokine levels at the end of the active condition compared to the beginning of the block, along with no statistical change at the end of the sham block condition compared to the beginning of the sham block, may indicate a more ideal treatment outcome.
Effects of PBMT versus Sham PBMT on Saliva Biomarkers | Through study completion, an average of 8 weeks.
  Changes in saliva biomarkers (cytokine panel: IL-1 Beta, IL-6, IL-8 & TNF-alpha) compared across the sham and active PBMT conditions. As elevated proinflammatory cytokines may be a sign of heightened inflammation, lower cytokine levels in saliva samples at the end of the active condition compared to the beginning of the block, along with no statistical change at the end of the sham block condition compared to the beginning of the sham block, may indicate a more ideal treatment outcome.
Effects of PBMT versus Sham PBMT on Heart Rate | Through study completion, an average of 8 weeks.
  Acute heart rate variability differences within a single treatment session and trends across treatment weeks compared to sham PBMT. Higher heart rate variability and/or lower resting heart rate during active PBMT may indicate a more ideal treatment outcome.
Effects of PBMT versus Sham PBMT on Defense Veterans Pain Rating Scale Scores | Through study completion, an average of 8 weeks.
  Differences in self reported Defense Veterans Pain Rating Scale (DVPRS) scores during active PBMT weeks are compared with baseline and sham PBMT weeks. The Defense Veterans Pain Rating Scale is a 0-10 color coded scale where green represents mild pain with a scale ranging from 0-4; yellow represents moderate pain with a scale ranging from 5-6, and red represents severe pain with a scale ranging from 7-10. Lower DVPRS scores in active PBMT conditions when compared to sham conditions would indicate a more ideal treatment outcome.
Effects of PBMT versus Sham PBMT on Athletic Mental Energy Scale Scores | Through study completion, an average of 8 weeks.
  Differences in self reported Athletic Mental Energy Scale (AMES) scores during active PBMT weeks are compared with baseline and sham PBMT weeks. The Athletic Mental Energy Scale comprises 18 items measuring athletes' perception of their energy state, including vigor, confidence, motivation, tirelessness, concentration, and calm. Participants rate their feelings on a 6-point Likert scale (1 = not at all, 6 = completely so). Higher AMES scores in active PBMT conditions when compared to sham conditions could indicate a more ideal treatment outcome.
Effects of PBMT versus Sham PBMT on Epworth Sleepiness Scale Scores | Through study completion, an average of 8 weeks.
  Differences in self reported Epworth Sleepiness Scale scores during active PBMT weeks are compared with baseline and sham PBMT weeks. The Epworth Sleepiness Scale results range from 0 to 24. Results from 0 to 10 show average (normal) daytime sleepiness, results under 10 may not be cause for concern or could identify trouble sleeping (insomnia), 11 to 24 indicates excessive (abnormal) daytime sleepiness. Lower Epworth Sleepiness Scale Scores scores in active PBMT conditions when compared to sham conditions could indicate a more ideal treatment outcome.

SECONDARY OUTCOMES:
Effects of using PBMT Light Beds at Different Power Intensities on Anti-Inflammatory Blood Biomarkers | Through study completion, an average of 8 weeks.
  Changes in blood biomarkers (MSD anti-inflammatory panel: IL-4, IL-10) compared across low-power and high-power PBMT. As elevated anti-inflammatory cytokine levels may be a sign of lowered inflammation, higher anti-inflammatory cytokine levels may indicate a more ideal treatment outcome.
Effects of using PBMT Light Beds at Different Power Intensities on Proinflammatory Blood Biomarkers | Through study completion, an average of 8 weeks.
  Changes in blood biomarkers (MSD proinflammatory panel: IL-1beta, IL-2, IL-6, IL-12p70, IL-17A, IFN-gamma, and TNF-alpha) compared across low-power and high-power PBMT. As elevated proinflammatory cytokine levels may be a sign of heightened inflammation, lower proinflammatory cytokine levels may indicate a more ideal treatment outcome.
Effects of using PBMT Light Beds at Different Power Intensities on Saliva Biomarkers | Through study completion, an average of 8 weeks.
  Changes in saliva biomarkers (cytokine panel: IL-1 Beta, IL-6, IL-8 & TNF-alpha) compared across high-power and low-power PBMT. As elevated proinflammatory cytokines may be a sign of heightened inflammation, lower cytokine levels in saliva samples may indicate a more ideal treatment outcome.
Effects of using PBMT Light Beds at Different Power Intensities on Heart Rate | Through study completion, an average of 8 weeks.
  Acute heart rate variability differences within a single treatment session and trends across treatment weeks compared across low-power and high-power PBMT treatment.
Effects of using PBMT Light Beds at Different Power Intensities on Defense Veterans Pain Rating Scale Scores | Through study completion, an average of 8 weeks.
  Differences in self reported Defense Veterans Pain Rating Scale scores compared across low-power and high-power PBMT treatment. The Defense Veterans Pain Rating Scale is a 0-10 color coded scale where green represents mild pain with a scale ranging from 0-4; yellow represents moderate pain with a scale ranging from 5-6, and red represents severe pain with a scale ranging from 7-10.
Effects of using PBMT Light Beds at Different Power Intensities on Athletic Mental Energy Scale Scores | Through study completion, an average of 8 weeks.
  Differences in self reported Athletic Mental Energy Scale scores compared across low-power and high-power PBMT treatment. The Athletic Mental Energy Scale comprises 18 items measuring athletes' perception of their energy state, including vigor, confidence, motivation, tirelessness, concentration, and calm. Participants rate their feelings on a 6-point Likert scale (1 = not at all, 6 = completely so).
Effects of using PBMT Light Beds at Different Power Intensities on Epworth Sleepiness Scale Scores | Through study completion, an average of 8 weeks.
  Differences in self reported Epworth Sleepiness Scale scores compared across low-power and high-power PBMT treatment. The Epworth Sleepiness Scale results range from 0 to 24. Results from 0 to 10 show average (normal) daytime sleepiness, results under 10 may not be cause for concern or could identify trouble sleeping (insomnia), 11 to 24 indicates excessive (abnormal) daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Eckerle, Principal Investigator — United States Air Force Research Laboratory
Locations (1):
- Wright Patterson Air Force Base, Beavercreek, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ailioaie LM, Litscher G. Photobiomodulation and Sports: Results of a Narrative Review. Life (Basel). 2021 Dec 3;11(12):1339. doi: 10.3390/life11121339. PMID 34947870
- [Background] Anders JJ, Lanzafame RJ, Arany PR. Low-level light/laser therapy versus photobiomodulation therapy. Photomed Laser Surg. 2015 Apr;33(4):183-4. doi: 10.1089/pho.2015.9848. No abstract available. PMID 25844681
- [Background] Heiskanen V, Hamblin MR. Photobiomodulation: lasers vs. light emitting diodes? Photochem Photobiol Sci. 2018 Aug 8;17(8):1003-1017. doi: 10.1039/c8pp90049c. PMID 30044464
- [Background] Rossato M, Dellagrana RA, Sakugawa RL, Baroni BM, Diefenthaeler F. Dose-Response Effect of Photobiomodulation Therapy on Muscle Performance and Fatigue During a Multiple-Set Knee Extension Exercise: A Randomized, Crossover, Double-Blind Placebo-Controlled Trial. Photobiomodul Photomed Laser Surg. 2020 Dec;38(12):758-765. doi: 10.1089/photob.2020.4820. Epub 2020 Nov 24. PMID 33232629
- [Background] Tumilty S, Mani R, Baxter GD. Photobiomodulation and eccentric exercise for Achilles tendinopathy: a randomized controlled trial. Lasers Med Sci. 2016 Jan;31(1):127-35. doi: 10.1007/s10103-015-1840-4. Epub 2015 Nov 26. PMID 26610637
- [Background] de Paiva PR, Tomazoni SS, Johnson DS, Vanin AA, Albuquerque-Pontes GM, Machado CD, Casalechi HL, de Carvalho PT, Leal-Junior EC. Photobiomodulation therapy (PBMT) and/or cryotherapy in skeletal muscle restitution, what is better? A randomized, double-blinded, placebo-controlled clinical trial. Lasers Med Sci. 2016 Dec;31(9):1925-1933. doi: 10.1007/s10103-016-2071-z. Epub 2016 Sep 13. PMID 27624781

DOCUMENTS (1):
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT06403644/ICF_000.pdf